CLINICAL TRIAL: NCT02161952
Title: Pirfenidone, an Antifibrotic and Antiinflammatory Drug for Treatment of Patients With Cirrhosis Due to Hepatitis C Virus. Phase II/III Study
Brief Title: Pirfenidone, an Antifibrotic and Antiinflammatory Drug
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Collaborators: Cell Therapy And Technology, S.a. De C.v. (Industry)
Responsible Party: Principal Investigator, Juan Armendáriz-Borunda, Head, Molecular Biology and Genomics Department, CUCS, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IBMMTG.05; HCG, No. Registry 505/05 (Registry Identifier: COFEPRIS, No. Registry 05330020020126)
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-06

CONDITIONS: Fibrosis; Hepatitis C Chronic
Keywords: Fibrosis, necroinflammation, hepatitis C chronic
MeSH Terms: conditions — Fibrosis; Hepatitis C, Chronic | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pirfenidone (Experimental): Pirfenidone 400 mg capsules, orally administered thrice daily to yield a daily dose of 1200 mg during two years.
  Interventions: Drug: Pirfenidone
- Matched equivalent placebo (Placebo Comparator): Matched equivalent placebo
  Interventions: Drug: Matched equivalent placebo

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone was supplied orally in 400 mg gel capsules three times daily (every 8 hours) for a full dosage of 1200 mg daily during 24 months.
  Other Names: 5 methyl-1-phenil-2 (1H)-pyridone
  Arms: Pirfenidone
Drug: Matched equivalent placebo
  Arms: Matched equivalent placebo

SUMMARY:
The aim of this study was to assess whether two-year treatment with Pirfenidone influence necro-inflammation, fibrosis and steatosis in patients with chronic hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established advanced liver disease caused by hepatitis C virus (HCV) chronic infection defined by a positive test for anti-HCV antibodies and detectable serum HCV RNA (Amplicor HCV 2.0 polymerase chain reaction (PCR) assay).
* Sign an informed consent form to allow the collection of liver biopsies before and after treatment.
* No antifibrotic, antiviral or immunosuppressive drugs for at least 6 months before starting pirfenidone therapy.
* No alcohol intake for at least 6 months before nor during Pirfenidone (PFD) treatment.

Exclusion Criteria:

* Patients with clinical contraindications to hepatic biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-05; Primary Completion 2006-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Fibrosis staging | 24 months
  Fibrosis was evaluated according to Ishak fibrosis staging scale.

SECONDARY OUTCOMES:
Grade of necroinflammation activity | 24 months
  Necroinflammatory activity was evaluated according to the Ishak modified histological activity index (HAI).

CONTACTS AND LOCATIONS:
Overall Officials: Juan Armendariz-Borunda, Ph. D., Principal Investigator — Head, Molecular Biology and Genomics Department

REFERENCES:
- [Derived] Flores-Contreras L, Sandoval-Rodriguez AS, Mena-Enriquez MG, Lucano-Landeros S, Arellano-Olivera I, Alvarez-Alvarez A, Sanchez-Parada MG, Armendariz-Borunda J. Treatment with pirfenidone for two years decreases fibrosis, cytokine levels and enhances CB2 gene expression in patients with chronic hepatitis C. BMC Gastroenterol. 2014 Jul 27;14:131. doi: 10.1186/1471-230X-14-131. PMID 25064094